CLINICAL TRIAL: NCT04923919
Title: Clinical Study of Chimeric Antigen Receptor T Lymphocytes (CAR-T) in the Treatment of Myeloid Leukemia
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: 920th Hospital of Joint Logistics Support Force of People's Liberation Army of China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BG-CT-19-005
Record Dates: First submitted 2021-05-08; First posted 2021-06-11 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm (Experimental): CLL-1 targeting CAR-T treatment
  Interventions: Drug: Anti-CLL1 CART cells

INTERVENTIONS:
Drug: Anti-CLL1 CART cells — In this study, patients with acute myeloid leukemia were treated with autologous anti-CLL1 CAR T cells by a single, intravenous infusion.Blood and bone marrow were collected before and 12 months after infusion to detect the number and activity of CAR T cells, and to evaluate the efficacy of CAR T cells.
  Other Names: CLL1 CAR-T

SUMMARY:
Researchers plan to enroll a total of 100 patients with relapsed, refractory acute myeloid leukemia (AML) to receive a single dose of autologous CAR T cells.The safety of CAR T therapy was evaluated by observing adverse events after cell therapy;The efficacy of CAR-T therapy was evaluated against the outcome of patients' own past standard treatment regimens or historical data.Blood and bone marrow were collected before and 12 months after infusion to detect the number and activity of CAR T cells, and to evaluate the pharmacokinetics (PK) of CAR T cells.

ELIGIBILITY:
Inclusion Criteria:

1. The diagnosis of myeloid leukemia was clear;Refractory treatment was defined as: (1) 2 patients who did not achieve partial remission after treatment with standard induced remission regimens.② The patients who relapsed within 6 months after the first remission were also called early recurrence.③ The failure relapsed 6 months after the initial response, but was retreated with the original induced response regimen.(4) multiple relapse.Relapse is defined as: patients who achieve complete remission after treatment, more than 5% of leukemia cells in the bone marrow, also known as intramedullary recurrence;Or the presence of leukaemia outside the bone marrow, also known as extramedullary relapse (usually in the central nervous system, testicular leukemia is the most common);
2. Diseased cells were confirmed to express CD123, CLL1 and other targets;
3. KPS > 60 points;
4. Expected survival of more than 3 months;
5. No gender limitation, age 2-75;
6. Patients clinically diagnosed as high-risk type, refractory type of recurrence or not eligible for standard treatment;
7. No serious mental disorders;
8. Sufficient heart, liver and renal function (a. Liver function: ALT/AST < 3 times upper limit of normal value (ULN) and bilirubin ≤34.2μmol/L;B. Renal function: creatinine < 220μmol/L;C. Lung function: indoor oxygen saturation ≥95%;D. Cardiac function: left ventricular ejection fraction (LVEF) ≥40%;);
9. No other serious diseases (such as autoimmune diseases, immune deficiency, organ transplantation) that are in conflict with this program;
10. Can cooperate with trial management and follow-up;
11. Patients voluntarily participated in the study and signed the informed consent

Exclusion Criteria:

1. History of other malignant tumors;
2. Uncontrolled active infection;
3. Patients with underlying diseases requiring systemic use of glucocorticoids;
4. Acute or chronic GVHD;
5. T-cell inhibitor therapy;
6. Pregnant and lactating women;
7. Patients with active hepatitis B;
8. Other conditions considered by the investigator to be inappropriate for the study (HIV infection, intravenous drug addiction, etc.), or other conditions that may affect the analysis of the results of the clinical study.

Ages: 2 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-09-14 (Actual); Primary Completion 2024-12-05 (Estimated); Study Completion 2024-12-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of AE after CAR-T infusion | up to 12 months after CAR-T infusion
  Incidence of adverse events after CAR-T infusion
  Data. The records of adverse events (AE) should include: description of AE and all related symptoms, occurrence time, severity, duration, measures taken, final results and outcomes. According to NCI CTC AE 5.0 standard, AE was scored
  Grade.
  Safety evaluation indexes include but are not limited to the following contents
  1. Any spontaneously reported and all directly observed adverse events;
  2. Any abnormal changes in vital signs and physical examination;
  3. The abnormal results of laboratory examination, physical examination and blood examination with clinical significance after treatment

SECONDARY OUTCOMES:
ORR rate | 1month, 2 months, 3months, 6months ,12months after CAR-T infusion
  Overall response rate (ORR=CR+CRi) after CAR-T infusion
PFS | 1month, 2 months, 3months, 6months ,12months after CAR-T infusion
  Progression free survival (PFS) after CAR-T infusion
OS | 1month, 2 months, 3months, 6months ,12months after CAR-T infusion
  overall survival (OS) after CAR-T infusion
Change of CAR Copies | Days 4, 7, 10, 14 and months 2, 3, 6, 9, 12 after Fast Dual CAR-T infusion
  CAR Copies measured by qPCR after CAR-T infusion
Change of CAR-T cell counts | Days 4, 7, 10, 14 and months 2, 3, 6, 9, 12 after Fast Dual CAR-T infusion
  CAR-T cell counts measured by Flow cytometry after CAR-T infusion

CONTACTS AND LOCATIONS:
Locations (1):
- No.212 Daguan Road, Xishan District, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: No